CLINICAL TRIAL: NCT00601549
Title: A Randomized Controlled Clinical Trial Comparing Oncological Results and Functional Recovery Between Laparoscopic and Open Method for the Treatment of Advanced Rectal Cancer After Concurrent Chemoradiation Therapy (CCRT)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 941007; NSC96-2314-B-002-146
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; CCRT; Laparoscopic Surgery; rectal cancer can be resected by curative and elective surgery; rectal adenocarcinoma below peritoneal reflection; American Society of Anesthesiology（ASA） classⅠ to Ⅲ lesions
MeSH Terms: conditions — Rectal Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients with low rectal cancer after CCRT undergoing laparoscopic surgery
  Interventions: Procedure: Laparoscopic surgery
- 2 (Active Comparator): Patients with low rectal cancer after CCRT undergoing traditional open surgery
  Interventions: Procedure: Traditional open surgery

INTERVENTIONS:
Procedure: Laparoscopic surgery — Laparoscopic surgery
  Arms: 1
Procedure: Traditional open surgery — Open surgery
  Arms: 2

SUMMARY:
This is a three-year research project. The major aims of this study are to:(1) compare the functional recovery and oncologic results in patients with advance rectal cancer treated by either traditional open or laparoscopic methods by randomized prospective clinical trials;(2) investigate the presence of tumor cells in the peripheral blood of patients undergoing either laparoscopic or open surgery; (3) searching for the clinicopathologic features of advanced rectal cancer after CCRT; (4) conduct the translational research regarding the difference of gene expression and its prognostic significance in advanced rectal cancer before and after chemoradiation therapy by micro-array analysis methods; (5) exploration of the potential stem cells of colorectal cancer using CD-133 cell surface marker.

DETAILED DESCRIPTION:
With the progress of medical technology, the minimally invasive laparoscopic colorectal surgery is currently enthusiastically performed in the medical center all over the world. Because preoperative CCRT can induce fibrosis of pelvic tissues, most colorectal surgeons have been hesistant to apply the laparoscopic approach to the resection of irradiated rectal cancer. However, based on our preliminary experience(Liang et al. Dis Colon Rectum Sep,2005), we found that if rectal cancers were resected by laparoscopic approach, the advantages include better visualization of anatomical structures such as paired hypogastric nerves, presacral fascia, lateral ligament, seminal vesicles and middle hemorrhoidal artery, as compared to traditional open method. Moreover, the conduction of laparoscopic double-stapling technique or pull-through procedure was not jeopardized by CCRT even when the pelvis is narrow in male patient. That is, with the current surgical technique, we feel that laparoscopic procedure is feasible and safe for inrradiated rectal cancers. Because the application of this technique in the resection of rectal cancer after CCRT is not reported before and has academic importance, it is mandatory for us to conduct this randomized prospective study. Remarkably, some objective surgical stress-related factors including CD4+/CD8+, ESR, CRP, and IL-6 (both in serum and intra-peritoneal surgical wounds), and the presence of cancer cells in either laparoscopic and open group of patients were analyzed and compared. Moreover, the translational research regarding the expression of genes and their prognostic significance before and after chemoradiation therapy have been scarce. In this project, we plan to explore the influence of chemo radiation therapy on the gene expression by microarray analysis according to the reproducible experiences developed by our colleagues in the research of gastric cancer (JCO 2005;23:7286-95). Initially, we will focus on the expression difference of the commonly mentioned genes related to the chemosensitivity of colorectal cancer, including mismatch repair genes, thymidylate synthetase, Dipyrimidine dehydrogenase (DPD), and epidermal growth factor receptor (EGFR), and then extend to the screening of the whole genome. Moreover, some recent reports indicated that the cell population harboring CD-133 were ther potential colorectal cancer stem cells. In this project, we will also explore the changes of histopathology and CD-133 cellular population in advanced rectal cancer after CCRT.

Because this is a randomized prospective clinical trial, it is uneasy to accrue enough patients. According to the statistical estimation, at least 558 patients should be recruited and randomized to either traditional open group and laparoscopic group to reach a statistical significance. Moreover, it has been reported that in order to represent the overall survival, the patients have to be followed up for at least 3 years after treatment. Therefore, it is necessary that this project should be further conducted for at least 3 years. Based on our preliminary results in the previous 2-year conduction of this project, we found that laparoscopic technique facilitated patients with rectal cancer after CCRT less surgical invasiveness, faster postoperative recovery, similar extent of dissection and the number of harvested lymph nodes, and did not increase of tumor dissemination during surgical manipulation, as compared with traditional open surgery. This encouraging results inspired us to complete this 3-year project, with a view to enhancing the academic reputation of Taiwan Colorectal Surgery and the quality of clinical management for patients with rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer can be resected by curative and elective surgery.
* Rectal adenocarcinoma below peritoneal reflection
* American Society of Anesthesiology（ASA） classⅠ to Ⅲ lesions

Exclusion Criteria:

* Cancer located at upper rectum （above peritoneal reflection）
* Distant metastasis
* Adjacent organ invasion
* Intestinal obstruction
* Past colonic surgery
* Body mass index（BMI）>35 kg/m2
* Patients who can not complete the whole treatment protocol of concurrent chemoradiation therapy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2000-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Oncologic Results | Every 6 months

SECONDARY OUTCOMES:
Functional recovery of patients | every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tung Liang, PhD, Principal Investigator — Division of Colorectal Surgery, Department of Surgery , National Taiwan University Hospital
Locations (1):
- Division of Colorectal Surgery, Department of Surgery , National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Liang JT, Huang KC, Lai HS, Lee PH, Jeng YM. Oncologic results of laparoscopic versus conventional open surgery for stage II or III left-sided colon cancers: a randomized controlled trial. Ann Surg Oncol. 2007 Jan;14(1):109-17. doi: 10.1245/s10434-006-9135-4. Epub 2006 Oct 25. PMID 17066227